CLINICAL TRIAL: NCT00005032
Title: A Phase I/II Study of G3139, a BCL-2 Antisense Oligonucleotide, Combined With Paclitaxel for the Treatment of Recurrent Small Cell Lung Cancer
Brief Title: Bcl-2 Antisense Oligodeoxynucleotide G3139 and Paclitaxel in Treating Patients With Recurrent Small Cell Lung Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Chicago (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10117; UCCRC-10017; NCI-T98-0091
Record Dates: First submitted 2000-04-06; First posted 2004-06-04 (Estimated); Last update posted 2013-02-11 (Estimated); Status verified 2013-02

CONDITIONS: Lung Cancer
Keywords: recurrent small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Small Cell Lung Carcinoma | interventions — oblimersen; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm A (Experimental): G3139 (3 mg/kg/day continuous IV infusion over 7 days every 21 days), Paclitaxel (150 mg/m2, 3 hr IV infusion on Day 6 of every 21 day cycle)
  Interventions: Biological: oblimersen sodium; Drug: paclitaxel

INTERVENTIONS:
Biological: oblimersen sodium
Drug: paclitaxel

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Bcl-2 antisense oligodeoxynucleotide G3139 may increase the effectiveness of a chemotherapy drug by making tumor cells more sensitive to the drug.

PURPOSE: Phase I/II trial to study the effectiveness of bcl-2 antisense oligodeoxynucleotide G3139 and paclitaxel in treating patients who have recurrent small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Assess the toxicity and feasibility of paclitaxel administration during continuous intravenous bcl-2 antisense oligodeoxynucleotide G3139 in patients with recurrent small cell lung cancer. II. Evaluate the clinical response of this patient population when treated with this regimen. III. Evaluate the correlation between bcl-2 expression in these patients and efficacy of this therapy.

OUTLINE: Patients are stratified according to whether they have received prior taxane therapy (yes vs no). Patients receive bcl-2 antisense oligodeoxynucleotide G3139 IV continuously on days 1-6 followed by 2 weeks of rest. Paclitaxel IV is administered over 3 hours on day 6 of each course. Treatment continues for a minimum of 2 courses in the absence of disease progression or unacceptable toxicity. Intrapatient dose escalation is allowed. Patients are followed until death.

PROJECTED ACCRUAL: A total of 19-33 patients will be accrued for this study within 12-18 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically or cytologically confirmed small cell lung cancer Prior therapy including either cisplatin or carboplatin with progression either on therapy or within 3 months of completing therapy Bidimensionally measurable disease on CT scan or x-ray, not limited to the CNS No active CNS disease CNS metastasis allowed if measurable disease outside of CNS and completed a course of CNS radiotherapy if clinically indicated and recovered

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: ECOG 0-2 OR Zubrod 0-2 Life expectancy: Not specified Hematopoietic: WBC at least 3,000/mm3 Hemoglobin at least 9 g/dL Platelet count at least 100,000/mm3 Hepatic: Bilirubin no greater than 1.5 mg/dL ALT/AST no greater than 2 times upper limit of normal (ULN) Alkaline phosphatase no greater than 2 times ULN Renal: Creatinine no greater than 1.5 mg/dL OR Creatinine clearance at least 50 mL/min Cardiovascular: No evidence of heart block greater than first degree, bundle branch block, or ventricular or supraventricular arrhythmia on EKG No clinical evidence of congestive heart failure, angina, or documented myocardial infarction within past 6 months Other: Not pregnant or nursing Negative pregnancy test Fertile patients must use effective contraception No known hypersensitivity to Cremaphor EL No other significant concurrent medical or psychiatric condition that might place patient at increased risk from study

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: See Disease Characteristics Endocrine therapy: Not specified Radiotherapy: See Disease Characteristics At least 4 weeks since prior radiotherapy to only site of measurable disease or to greater than 20% of bone marrow Surgery: Not specified Other: No other concurrent experimental drugs or cancer therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2000-04; Primary Completion 2001-01 (Actual); Study Completion 2001-09 (Actual)

PRIMARY OUTCOMES:
Tolerability of dosing | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Charles M. Rudin, MD, PhD, Study Chair — University of Chicago
Locations (11):
- United States (11):
  - University of Illinois at Chicago, Chicago, Illinois
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - Louis A. Weiss Memorial Hospital, Chicago, Illinois
  - Cancer Care Specialists of Central Illinois, S.C., Decatur, Illinois
  - Evanston Northwestern Health Care, Evanston, Illinois
  - Division of Hematology/Oncology, Park Ridge, Illinois
  - Oncology/Hematology Associates of Central Illinois, P.C., Peoria, Illinois
  - Central Illinois Hematology Oncology Center, Springfield, Illinois
  - Fort Wayne Medical Oncology and Hematology, Inc., Fort Wayne, Indiana
  - Michiana Hematology/Oncology P.C., South Bend, Indiana
  - Arthur G. James Cancer Hospital - Ohio State University, Columbus, Ohio

REFERENCES:
- [Result] Rudin CM, Otterson GA, Mauer AM, Villalona-Calero MA, Tomek R, Prange B, George CM, Szeto L, Vokes EE. A pilot trial of G3139, a bcl-2 antisense oligonucleotide, and paclitaxel in patients with chemorefractory small-cell lung cancer. Ann Oncol. 2002 Apr;13(4):539-45. doi: 10.1093/annonc/mdf124. PMID 12056703